CLINICAL TRIAL: NCT04061447
Title: Tailored Antibiotic Susceptibility-guided Therapy Via Gastric Juice PCR for First-line H Pylori Eradication, a Prospective Randomized Controlled Trial
Brief Title: Tailored Juice-guided Eradication Therapy
Acronym: HP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University (Other)
Responsible Party: Principal Investigator, DENG-CHYANG WU, Clinical Professor, Kaohsiung Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KMUHIRB-G(I)-20150043
Record Dates: First submitted 2019-08-16; First posted 2019-08-19 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2016-02

CONDITIONS: Helicobacter Pylori Infection
Keywords: gastric juice guided therapy; H.pylori eradication

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- susceptibility-guided therapy (Experimental): In the group of the empirical triple therapy, patients received rabeprazole 20mg B.I.D, amoxicillin 1000mg B.I.D, and clarithromycin 500mg B.I.D for seven days.
  Interventions: Drug: susceptibility-guided therapy
- empirical clarithromycin-based triple therapy (Active Comparator): In the group of gastric juice susceptibility-guided therapy, the eradication regimen was based on the susceptibility results of gastric PCR. If clarithromycin was sensitive, the regimen contained rabeprazole 20mg B.I.D, amoxicillin 1000mg B.I.D, and clarithromycin 500mg B.I.D for seven days. If clarithromycin was resistant and levofloxacin was sensitive, the regimen was rabeprazole 20mg B.I.D, amoxicillin 1000mg B.I.D, and levofloxacin 500mg QD for seven days. If clarithromycin and levofloxacin were both resistant, the regimen was either reverse-hybrid therapy (rabeprazole 20mg B.I.D x 14 days, amoxicillin 1000mg B.I.D, x 14 days, clarithromycin 500mg B.I.D for 7 days, and metronidazole 500mg B.I.D for 7 days) or high dose dual therapy (rabeprazole 20mg Q.I.D and amoxicillin 1000mg Q.I.D for 14 days). Owing to this open design, either reverse-hybrid therapy or high dose dual therapy was chosen by doctors' preference.
  Interventions: Drug: empirical clarithromycin-based triple therapy

INTERVENTIONS:
Drug: susceptibility-guided therapy — rabeprazole 20mg B.I.D, amoxicillin 1000mg B.I.D, and clarithromycin 500mg B.I.D for seven days.
  Arms: susceptibility-guided therapy
Drug: empirical clarithromycin-based triple therapy — The eradication regimen was based on the susceptibility results of gastric PCR. If clarithromycin was sensitive, the regimen contained rabeprazole 20mg B.I.D, amoxicillin 1000mg B.I.D, and clarithromycin 500mg B.I.D for seven days. If clarithromycin was resistant and levofloxacin was sensitive, the regimen was rabeprazole 20mg B.I.D, amoxicillin 1000mg B.I.D, and levofloxacin 500mg QD for seven days. If clarithromycin and levofloxacin were both resistant, the regimen was either reverse-hybrid therapy (rabeprazole 20mg B.I.D x 14 days, amoxicillin 1000mg B.I.D, x 14 days, clarithromycin 500mg B.I.D for 7 days, and metronidazole 500mg B.I.D for 7 days) or high dose dual therapy (rabeprazole 20mg Q.I.D and amoxicillin 1000mg Q.I.D for 14 days). Owing to this open design, either reverse-hybrid therapy or high dose dual therapy was chosen by doctors' preference.
  Arms: empirical clarithromycin-based triple therapy

SUMMARY:
In this study, the investigators aim to investigate the efficacy of tailored anti-microbial susceptibility guided-therapy via gastric juice PCR, compared with empirical standard triple therapy.

DETAILED DESCRIPTION:
The eradication of H. pylori is an important clinical issue due to its association with many gastrointestinal diseases such as peptic ulcer and even gastric cancer. However, with the global trend of increasing antibiotic resistance, the eradication rate of clarithromycin-based standard triple therapy has declined to less than 80%. To overcome such alarming antibiotic resistance, antimicrobial susceptibility-guided therapy is recommended. However, the literature on gastric juice PCR as susceptibility-guided therapy is scant; therefore, the investigators conducted this prospective randomized controlled trial with the aim of investigating the efficacy of antibiotic susceptibility-guided therapy via gastric juice PCR for first-line eradication.

ELIGIBILITY:
Inclusion Criteria:

1. male or non-pregnant female aged more than 20 yeasrs
2. H.pylori infection
3. Mental and legal ability to give a written infomed consent

Exclusion Criteria:

1. pregnant women
2. previous allergic reaction to antibiotics (clarithromycin, amoxicillin, levofloxacin, metronidazole and Proton-pump inhibitor(rabeprazole)
3. patients with previous gastric surgery
4. the coexistence of serious concomitant illness(for example, decompensated liver cirrhosis, uremia)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2016-02-05 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
The rate of H.pylori eradication | 6 weeks
  Four-to-six weeks after treatment, all patients received the 13C-urea breath test to confirm H. pylori infection status.

CONTACTS AND LOCATIONS:
Overall Officials: Deng-Chyang Wu, MD, PHD, Study Chair — Kaohsiung Medical University; Chao-Hung Kuo, MD, PHD, Principal Investigator — Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No